CLINICAL TRIAL: NCT00069914
Title: Immune Response to Influenza Vaccination in HIV-Infected Individuals
Brief Title: Immune Response to Influenza Vaccine in HIV-Infected Individuals
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030310; 03-I-0310
Record Dates: First submitted 2003-10-02; First posted 2003-10-03 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: Immunization; Immune Activation; Flu; Antibodies; Titers; HIV; Healthy Volunteer; HV
MeSH Terms: conditions — HIV Infections; Influenza, Human

SUMMARY:
This study will evaluate how HIV infection, including CD4 cell count and viral load, affects the patient's ability to produce antibodies in response to vaccination with the influenza (flu) vaccine. Earlier studies have shown that people with HIV infection do not respond as well as healthy subjects to flu vaccine; that is, they don't make as many antibodies in response to the vaccine. Before the use of current anti-HIV medications, antibodies made to flu vaccination in HIV-positive individuals was related to their CD4 cell count. This trial will examine how CD4 counts and the amount of virus in the blood affect how much and what kind of antibodies the body makes to the flu vaccine.

HIV-infected patients and healthy normal volunteers between 18 and 60 years of age may be eligible for this study. Healthy subjects will serve as controls to make sure the flu vaccine works (i.e., stimulates production of enough antibody to protect against the flu), and to compare the amount of antibodies made by HIV-positive and HIV-negative people. Candidates will be screened with a medical history and blood tests (see below). Women who are able to have children will have a pregnancy test. Pregnant women are excluded from the study.

Participants will undergo the following procedures:

1. Blood drawing for the following tests:

   * Routine tests (complete blood count, kidney and liver functions, electrolyte levels).
   * CD4 cell count.
   * HLA typing (a genetic marker of the immune system) if it has not already been done at the NIH. This test may be used to try to identify factors associated with the rate of progression of HIV disease or related conditions. Determining HLA type is necessary to be able to perform certain research studies. Some HLA types have been associated with an increased risk of certain diseases like arthritis and other rheumatologic problems.
   * Viral load (HIV-infected patients only).
   * Influenza antibody levels.
   * B cell levels.
2. Flu vaccination
3. Follow-up visits on days, 7, 28, and 54 after vaccination for the following:

   * Review of any illnesses or fever.
   * Review of medications, if any changes were made.
   * Repeat blood tests.

DETAILED DESCRIPTION:
The purpose of this protocol is to evaluate the effect of HIV viral load and CD4 counts on the generation of influenza-specific antibodies and influenza-specific B cell responses in HIV-infected adults. HIV-infected subjects will be enrolled to receive the influenza vaccine appropriate to the on-going USA influenza season (Oct-March). Laboratory studies (including influenza titers, influenza-specific B cell frequencies, CD4 counts, and HIV viral loads) will be obtained at baseline (day of vaccination), day 7, 28, and 54 post-vaccination. HIV-negative healthy volunteers will serve as controls. Although there are some risks to influenza vaccine, the CDC Advisory Committee on Immunizations recommends influenza vaccination for HIV-infected patients. The primary study risks are those of phlebotomy and the inconvenience of multiple visits. Subjects will be compensated for participation in the study. Total enrollment of the study is a maximum of 165 subjects (132 HIV-infected individuals and 33 HIV-negative controls).

ELIGIBILITY:
INCLUSION CRITERIA:

HIV Positive:

1. Age greater than or equal 18 but less than or equal to 60 years old and willing and able to give informed consent
2. Enrollment during the USA influenza season (October-March)
3. Self-reported history of HIV infection at enrollment (If NIH HIV testing does not confirm that the subject is HIV-positive, the subject will be discontinued from the study and not included in the analysis.)

HIV Negative:

1. Age greater than or equal to 18 but less than or equal to 60 years old and willing and able to give informed consent
2. Enrollment during USA influenza season (October-March)
3. Self-reported healthy HIV-negative (If NIH HIV testing does not confirm that the subject is HIV-negative, the subject will be discontinued from the study and not included in the analysis.)

EXCLUSION CRITERIA:

HIV Positive:

1. Self-reported history of vaccination with the trivalent influenza preparation used for the current influenza season
2. Self-reported vaccination with any vaccine within the one month period prior to study enrollment
3. Acute febrile illness (may defer vaccine until resolved)
4. History of hypersensitivity to any influenza vaccine components including thimerosal or egg
5. History of Guillain-Barre syndrome
6. Intention to receive any other vaccine during the study period
7. Pregnancy
8. Self-reported treatment with immunomodulator/immunosuppressive drugs (interleukins, corticosteroids, or G(M)-CSF in the 4 weeks prior to enrollment
9. Self-reported history of IL-2 administration within the past 5 years
10. Use of theophylline preparations or warfarin because of the theoretical possibilities, of enhanced drug effects and toxicities post influenza vaccination
11. Active infection or other serious illness other than HIV that might affect the immune response to a vaccine
12. Current alcohol, substance abuse, or systemic/psychiatric illness that potentially could interfere with patient compliance and ability to make study visits

HIV Negative:

1. Self-reported history of vaccination with the trivalent influenza preparation used for the current influenza season
2. Self-reported vaccination with any vaccine within the one month period prior to study enrollment
3. Acute febrile illness (may defer vaccine until resolved)
4. History of hypersensitivity to any influenza vaccine components including thimerosal or egg
5. History of Guillain-Barre syndrome
6. Intention to receive any other vaccine during the study period
7. Pregnancy
8. Self-reported treatment with immunomodulator/immunosuppressive drugs (interleukins, corticosteroids, or G(M)-CSF in the 4 weeks prior to enrollment
9. Use of theophylline preparations or warfarin because of the theoretical possibilities, of enhanced drug effects and toxicities post influenza vaccination
10. Any medical conditions, or medication use might affect the immune response to a vaccine
11. Current alcohol, substance abuse, or systemic/psychiatric illness that potentially could interfere with patient compliance and ability to make study visit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 165
Dates: Start 2003-09; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] McNeil AC, Shupert WL, Iyasere CA, Hallahan CW, Mican JA, Davey RT Jr, Connors M. High-level HIV-1 viremia suppresses viral antigen-specific CD4(+) T cell proliferation. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13878-83. doi: 10.1073/pnas.251539598. PMID 11717444
- [Background] Moir S, Ogwaro KM, Malaspina A, Vasquez J, Donoghue ET, Hallahan CW, Liu S, Ehler LA, Planta MA, Kottilil S, Chun TW, Fauci AS. Perturbations in B cell responsiveness to CD4+ T cell help in HIV-infected individuals. Proc Natl Acad Sci U S A. 2003 May 13;100(10):6057-62. doi: 10.1073/pnas.0730819100. Epub 2003 May 1. PMID 12730375
- [Background] Kroon FP, van Dissel JT, de Jong JC, Zwinderman K, van Furth R. Antibody response after influenza vaccination in HIV-infected individuals: a consecutive 3-year study. Vaccine. 2000 Jul 1;18(26):3040-9. doi: 10.1016/s0264-410x(00)00079-7. PMID 10825608